CLINICAL TRIAL: NCT05467540
Title: Clinical Study of Spinery® A Novel Radio-Frequency Tumor Ablation Device for Spine Metastatic Tumors
Brief Title: Spinery® A Novel Radio-Frequency Tumor Ablation Device for Spine Metastatic Tumors
Acronym: SPARTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axon srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #2020-01
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Vertebral Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, no control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinery® RF Ablation System Arm (Experimental): Participants in this single-arm study underwent percutaneous radiofrequency ablation of painful bone metastases using the Spinery System, consisting of the Spinery® RF Generator, the sterile single-use Spinery® Kit, and the sterile single-use Spinery® Cooling Connection. The procedure was performed according to the study protocol, with follow-up visits scheduled at 1, 3, and 12 months to assess pain reduction, safety, usability, and quality of life.
  Interventions: Device: Spinery System

INTERVENTIONS:
Device: Spinery System — Radiofrequency ablation of bone metastases performed with the Spinery System, a radiofrequency generator with dedicated sterile, single-use accessories (electrode kit and cooling connection).
  Other Names: Spinery® RF Generator, the sterile single-use Spinery® Kit, and the sterile single-use Spinery® Cooling Connection

SUMMARY:
The SPARTA study (Spinery® Radiofrequency Ablation Device Study) is a prospective, multicenter, single-arm clinical investigation designed to evaluate the safety, performance, and efficacy of the Spinery® RF Generator and its sterile single-use accessories for the palliative treatment of painful bone metastases.

Adult patients with metastatic lesions involving the vertebral bodies, sacrum, iliac crest, or peri-acetabulum who were not candidates for, or had failed, standard therapies underwent percutaneous radiofrequency ablation with the investigational device.

A total of 52 participants were enrolled across five Italian centers and were assessed at baseline, post-procedure, and during follow-up visits at 1, 3, and 12 months.

Endpoints include evaluation of pain reduction, quality of life, usability, and procedural safety.

DETAILED DESCRIPTION:
Bone metastases are a frequent cause of pain and disability in patients with advanced cancer, often leading to impaired mobility and reduced quality of life. Conventional treatments such as systemic analgesics, radiotherapy, or chemotherapy may not always achieve adequate symptom control, particularly in patients with recurrent or resistant disease.

Radiofrequency (RF) ablation has emerged as a minimally invasive, image-guided procedure that induces controlled thermal necrosis within metastatic lesions, potentially reducing pain by interrupting nociceptive pathways and stabilizing the affected bone.

The SPARTA study was designed to collect clinical data on the Spinery® RF Generator and its sterile single-use accessories, a bipolar/monopolar RF ablation technology intended for percutaneous use in bone metastases.

This clinical investigation follows a prospective, multicenter, single-arm design without a control group; data are compared with published evidence available in the literature to contextualize safety and performance outcomes.

A total of 52 patients were enrolled across five Italian centers. Eligible participants were adults with painful metastatic bone tumors located in the thoracic or lumbar vertebrae, sacrum, iliac crest, or peri-acetabulum.

Following informed consent and baseline assessments, each patient underwent image-guided RF ablation using the Spinery® device. The procedure allowed the treating physician to select monopolar or bipolar cooled electrodes according to lesion size and location.

Participants were monitored within 24 hours post-procedure and followed at 1, 3, and 12 months after treatment.

Study assessments include:

* Pain evaluation using the Brief Pain Inventory (BPI)
* Quality of life assessment using the EQ-5D-5L questionnaire
* Functional performance using the Karnofsky Performance Scale
* Documentation of concomitant analgesic use and adverse events

The primary objectives are:

1. To evaluate short-term pain reduction at 3 months following treatment, as measured by changes in the BPI "worst pain" score.
2. To evaluate procedural safety, defined as the percentage of procedures completed without device-related adverse events, including nerve injury.

The secondary objectives are:

* To assess long-term pain reduction at 12 months.
* To evaluate usability and procedural performance (technical and procedural success without product-specialist intervention).
* To monitor quality-of-life and functional outcomes over the follow-up period.

This clinical investigation is conducted in compliance with ethical principles of Good Clinical Practice and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful metastatic malignant lesions involving bone;
* Patients, candidates to standard therapy, in which the RF ablation can be performed in combination with the Standard Therapy in accordance with the Investigator's indications;
* Patients who have failed, not candidates or refuse Standard Therapy (chemotherapy or radiotherapy);
* Patients with metastatic tumor size compatible with the expected ablation dimensions as reported for SPINERY devices in the IFU;
* Patients with localized pain resulting from not more than two sites of symptomatic metastatic disease
* Patients that do not have evidence of impending fracture
* Patients with metastatic lesions targeted for treatment located in the thoracic and/or lumbar vertebral body(ies), peri-acetabulum, iliac crest, and/or sacrum - no restrictions on location of lesion;
* Patients with BPI-Report worst pain score ≥4/10 at the target treatment site within the past 24 hours
* Patients with Karnofsky score ≥ 40 at enrollment
* Patients willing and able to provide a signed and dated informed consent, comply with the study plan, follow up visits and phone calls
* Patients at least 18 years old at the time of informed consent

Exclusion Criteria:

* Patients implanted with heart pacemaker or other implanted electronic device
* Patients with previous mechanical bone stabilization in the vertebral body to be treated
* Use of SPINERY in vertebral body levels C1-C7
* Multiple myeloma, solitary plasmacytoma, or primary malignant lesions in the index vertebra or bone.
* Active or incompletely treated local infection at the planned treatment site(s) and/or systemic infection.
* Planned treatment site(s) accompanied by objective evidence of secondary radiculopathy or neurologic compromise.
* Planned treatment site(s) associated with spinal cord compression or canal compromise requiring decompression.
* Fractures due to prostatic cancer or other osteoblastic metastases to the spine. Metastatic lesions originating in the prostate that are osteolytic or of mixed origin are eligible for the study.
* Pregnant, breastfeeding, or plan to become pregnant during the study duration.
* Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.
* Any condition that would interfere with the subject's ability to comply with study instructions or might confound the study interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Muto, Prof, MD, Study Director — Azienda Ospedaliera Antonio Cardarelli, Naples, Italy; Stefano Marini, MD, Principal Investigator — Ospedale Santissima Trinità, Cagliari, Italy; Francesco Amato, MD, Principal Investigator — Azienda Ospedaliera di Cosenza, Cosenza, Italy; Luigi Manfrè, MD, Principal Investigator — Istituto Oncologico del Mediterraneo, Catania, Italy; Matteo Bellini, MD, Principal Investigator — Azienda Ospedaliera Universitaria Senese, Siena, Italy
Locations (5):
- Italy (5):
  - Ospedale Santissima Trinità, Cagliari
  - Istituto Oncologico del Mediterraneo IOM, Catania
  - Azienda Ospedaliera di Cosenza, Cosenza
  - Azienda Ospedaliera Antonio Cardarelli, Naples
  - Azienda Ospedaliera Universitaria Senese, Siena

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between July 2022 and Nov 2023 at 5 clinical sites. Eligible participants were adult who met all inclusion/exclusion criteria specified in the protocol. Recruitment followed standard informed consent procedures at each site.
Pre-assignment Details: The Protocol Enrollment was 52 as planned. One participant withdrew consent after enrollment and prior to treatment allocation; therefore, 51 participants actually started the Spinery RF Ablation procedure. This explains the discrepancy between Protocol Enrollment and Started counts.
Groups:
- Spinery RF Ablation Treatment Group: This is a single-arm interventional group in which all enrolled patients receive treatment with the Spinery® RF Generator in combination with its sterile single-use accessories (Spinery® Kit and Spinery® Cooling Connection). The investigational device delivers bipolar cooled radiofrequency (RF) energy to spinal metastatic lesions with the objective of achieving thermal ablation of the tumor and palliative pain relief.
  Under image guidance (e.g., fluoroscopy or CT), one or two bipolar cooled probes are percutaneously inserted into the target lesion (vertebral bodies, sacrum, iliac crest, or peri-acetabulum). The RF ablation is performed with energy delivery up to 20 minutes per lesion, with optional cement injection. The treatment is intended for patients who failed, are not candidates for, or refuse standard therapy.
  This arm evaluates the safety, short-term (3 months) and long-term (12 months) efficacy of the RF treatment in reducing pain, as well as procedural performance and usability. All participants are assessed at baseline and followed up at 1, 3, 6, and 12 months.
Period: BaseLine
Arm/Group | Spinery RF Ablation Treatment Group
Started | 51
Completed | 51
Not Completed | 0
Period: 3-Month Follow-up
Arm/Group | Spinery RF Ablation Treatment Group
Started | 51
Completed | 41
Not Completed | 10
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Death | 5
Period: 12-Month Follow-up
Arm/Group | Spinery RF Ablation Treatment Group
Started | 41
Completed | 26
Not Completed | 15
Not completed — Lost to Follow-up | 6
Not completed — Death | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in all participants who started the Spinery RF Ablation procedure (N=51) prior to treatment. One participant withdrew consent after enrollment and before treatment allocation and was not included in the baseline analyses.
Groups:
- BaseLine: This single-arm group includes all patients enrolled and treated with the Spinery® RF Generator in combination with its sterile, single-use accessories (Spinery® Kit and Spinery® Cooling Connection). Each participant received radiofrequency (RF) ablation therapy targeted at bone metastatic lesions located in the vertebral bodies, sacrum, iliac crest, or peri-acetabulum. All procedures were image-guided and performed according to the protocol-defined treatment algorithm. Baseline demographic and clinical characteristics were collected before the ablation procedure and used to evaluate treatment efficacy and safety over time.
Arm/Group | BaseLine
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Primary Tumor Site [Number; unit: participants]
  Breast | 19
  Lungs | 12
  Prostate | 4
  Bladder | 1
  Kidney | 4
  Colon | 1
  Lynphatic system | 1
  Lymphomas | 1
  Sarcoma | 1
  Adeno Carcinoma | 1
  Intestine | 1
  Chest | 1
  Liver | 1
  Pancreas | 1
  Other | 1
Target Lesion Location [Count of Participants; unit: Participants]
  Vertebral Body | 27
  Sacrum | 10
  Iliac Crest | 7
  Pari-acetabulum | 7
Pain Score at Baseline (BPI) [Mean (Standard Deviation); unit: units on a scale] — Worst pain score at baseline was assessed using the Brief Pain Inventory (BPI), a validated scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Participants were asked to rate their worst pain in the last 24 hours prior to the RF ablation procedure. This measure was used to evaluate initial symptom severity and to assess changes in pain over time.
  units on a scale | 7.8 (1.6)
EQ-5D-5L [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life was assessed at baseline using the EQ-5D-5L questionnaire. The instrument evaluates five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) on five levels, scored from 1 (no problems) to 5 (extreme problems). Dimension scores can be combined using the EuroQol valuation set to calculate a single index value ranging from 0 (worst health state) to 90 (best health state). Higher scores indicate better health-related quality of life. This measure provides a standardized evaluation of baseline health status before treatment.
  units on a scale | 42.8 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worst Pain and Quality of Life Scores at 3 Months Using the Brief Pain Inventory (BPI) and EQ-5D-5L Questionnaires
Description: Pain severity and health-related quality of life were evaluated using two validated questionnaires:
  * Brief Pain Inventory (BPI): Participants rated their worst pain in the last 24 hours for each treated lesion site (thoracic, lumbar, peri-acetabulum, iliac crest, sacrum) on an 11-point numeric scale from 0 (no pain) to 10 (pain as bad as you can imagine).
  Higher scores indicate worse pain. The change in BPI Worst Pain Score was calculated as the average reduction from baseline to the 3-month visit.
  * EQ-5D-5L: Participants reported their overall health status across five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each rated on five levels of severity.
  Responses were converted into a utility index ranging from -0.594 (worst health state) to 1.000 (best health state), where higher scores indicate better quality of life.
  The EQ-5D-5L visual analogue scale (VAS) ranges from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: Baseline and 3-month follow-up
Population: All participants who started treatment and completed the 3-month follow-up visit are included in this analysis.
Measure: Mean (Standard Deviation); unit: points on a numeric scale
Groups:
- 3-Months Follow-up: This group includes all participants who completed the 3-month follow-up visit after Spinery RF Ablation treatment.
Arm/Group | 3-Months Follow-up
Number analyzed (Participants) | 41
points on a numeric scale
  Change in Worst Pain Score (BPI, 0-10 scale; higher = worse pain) | 3.4 (2.8)
  Change in Quality of Life (EQ-5D-5L VAS, 0-100 scale; higher = better health status) | 65.2 (19.0)

2. Primary Outcome: Number and Percentage of Participants Who Successfully Completed the Spinery® RF Ablation Procedure
Description: The number and percentage of participants who successfully completed the Spinery® RF ablation procedure per protocol.
  Completion is defined as participants who underwent the full planned treatment without premature discontinuation or technical interruption.
  Results are expressed as the count and percentage of the total number of treated participants.
Time Frame: Post-Procedure (primary evaluation point)
Population: All participants who started treatment and were evaluated for procedural completion.
Measure: Count of Participants; unit: Participants
Groups:
- Post-Procedure: This group includes all participants who underwent the Spinery® RF Ablation procedure. Outcome data collected at this time point include procedure completion and related immediate adverse events.
Arm/Group | Post-Procedure
Number analyzed (Participants) | 51
Participants | 51

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were assessed from the day of the Spinery® RF Ablation procedure through the 3-month follow-up visit. All-Cause Mortality was assessed from the day of the procedure through the 12-month follow-up visit.
Description: Serious and Other (Not Including Serious) Adverse Events were assessed from the day of the Spinery® RF Ablation procedure through the 3-month follow-up visit.
  All-Cause Mortality was assessed from the day of the procedure through the 12-month follow-up visit.
Groups:
- All Participants: This group includes all participants who underwent the Spinery® RF Ablation procedure with the Spinery® RF Generator and its sterile accessories. Adverse events were collected systematically at each clinical visit and via patient contact. Serious and non-serious procedure- or device-related adverse events were monitored from the day of the procedure through the 3-month follow-up visit. All-Cause Mortality was assessed from the day of the procedure through the 12-month follow-up visit. Events were evaluated for severity, seriousness, and relatedness to the procedure or device, in accordance with ISO 14155:2020. No modifications to standard AE/SAE definitions were applied.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 13/51
Serious Adverse Events (participants affected / at risk) | 13/51
Other Adverse Events (participants affected / at risk) | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=51)
Death (General disorders) | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=51)
New metastasis (right scapula) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Newly diagnosed right scapula metastasis occurring during follow-up, considered unrelated to the device or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT05467540/Prot_SAP_000.pdf